CLINICAL TRIAL: NCT01032824
Title: Community-based Self-management of HIV and Chronic Disease
Brief Title: Self-Managing HIV and Chronic Disease
Acronym: PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R01MH074380 (NIH)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: HIV/AIDS
Keywords: Complementary Therapies
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention (Experimental): Individual telephone counseling intervention.
  Interventions: Behavioral: Individual Telephone Counseling Intervention
- Group Arm (Other): Attention-matched comparison arm
  Interventions: Other: Group Arm
- Book Arm (Other): Information-matched control arm.
  Interventions: Other: Book Arm

INTERVENTIONS:
Behavioral: Individual Telephone Counseling Intervention — 10-session, 5-month HIV adherence and chronic disease self-management individual telephone counseling intervention.
  Other Names: telephone counseling
  Arms: Intervention
Other: Group Arm — 10-session didactic telephone group
  Other Names: Attention-matched comparison arm
  Arms: Group Arm
Other: Book Arm — Book only.
  Other Names: Information-matched comparison arm
  Arms: Book Arm

SUMMARY:
The purpose of this study is to conduct a randomized control trial of a behavioral intervention delivered by counselors via telephone to determine if this is an efficacious method for improving medication adherence and health-related quality of life for persons who are 50 and older and living with HIV/AIDS and other chronic conditions.

DETAILED DESCRIPTION:
450 adult HIV+ patients aged 50 or older will be randomized to one of three arms. 150 will be assigned to receive a series of ten 30-minute phone calls every two weeks from a counselor. 150 will be assigned to an attention-matched comparison arm, and will receive 10 sessions in a didactic telephone group. 150 will be assigned to a information-matched control arm and will receive the book Living Well with HIV & AIDS. Letters will be sent by AIDS Service Organizations inviting interested clients to call the study's 800 number to learn more about the study and to be screened for enrollment. Posters and brochures will also be posted in public areas of the ASOs. The individualized intervention combines problem-solving, with motivation and self-management. This trial will allow us to evaluate the effectiveness of a multi-component intervention on both specific HIV behavioral outcomes and non-disease-specific outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age 50 years or older
* HIV-positive serostatus
* currently prescribed antiretroviral medication
* antiretroviral nonadherence reported in past 30 days
* provision of oral informed consent

Exclusion Criteria:

* hearing problems that preclude participation in a telephone study
* presence of probable dementia or acute psychosis detectable by screening interview

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
antiretroviral (ART) adherence | Pre-treatment Screening and Baseline, 6, 9, and 12 months f/u.
health-related quality of life (physical, mental health, and social function) | Baseline, 6, 9, 12 mo f/u

SECONDARY OUTCOMES:
chronic disease treatment adherence | baseline, 6, 9 and 12 months f/u
Self-efficacy and readiness to change | baseline, 6, 9, 12 months f/u
perceived stress and depression | baseline, 6, 9, and 12 months f/u

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl L Catz, PhD, Principal Investigator — Group Health Research Institute
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States